CLINICAL TRIAL: NCT01223222
Title: A Randomised, Double-blind, Placebo-controlled, Phase IIa Pilot Study to Evaluate the Safety, Tolerability and Efficacy of Lytixar™ (LTX-109) in Patients With Uncomplicated, Gram-positive, Skin Infection
Brief Title: A Study to Evaluate Safety, Tolerability and Efficacy of Lytixar™ (LTX-109) on Uncomplicated, Gram-positive, Skin Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lytix Biopharma AS (Industry)
Responsible Party: Wenche Marie Olsen, Director of Development, Infectious Diseases, Lytix Biopharma AS
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10-109-03
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Gram-positive, Skin Infections; Mild Eczema/Dermatoses; Atopic Dermatitis
Keywords: Uncomplicated skin infections; Impetigo; Gram-negative; Diagnosis of uncomplicated, Gram-positive, skin infection. This may include patients with mild eczema/dermatoses such as atopic dermatitis.; Gram-positive organisms which in the opinion of the investigator are causative for infection of the lesion(s),
MeSH Terms: conditions — Cellulitis; Skin Diseases; Dermatitis, Atopic; Impetigo | interventions — L-arginyl-2,5,7-tris(1,1-dimethylethyl)-L-tryptophyl-N-(2-phenylethyl)-L-argininamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1% Lytixar™ (Placebo Comparator): 6 subjects will be treated with Lytixar™ and 2 will be treated with vehicle (placebo).
  Interventions: Drug: LTX-109
- 2% Lytixar™ (Active Comparator): 6 subjects will be treated with Lytixar™ and 2 will be treated with vehicle (placebo).
  Interventions: Drug: LTX-109
- 5% Lytixar™ (Active Comparator): 6 subjects will be treated with Lytixar™ and 2 will be treated with vehicle (placebo).
  Interventions: Drug: LTX-109

INTERVENTIONS:
Drug: LTX-109 — Topical administration. 3 times daily. 5 days.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Lytixar™ applied topically to uncomplicated skin infections.

Three dose levels of Lytixar™ (1%, 2% and 5%) versus placebo will be tested.

DETAILED DESCRIPTION:
Treatment of uncomplicated, Gram-positive, skin infection may include application of antiseptics and desiccants, but most importantly topical antibiotics. Guidance on the use of antimicrobial therapies has been published, poor prescribing practices still exist which facilitate the development of bacterial strains resistant to available therapy. The issue of antimicrobial resistance is particularly important for Gram-positive cocci such as Staphylococcus aureus and Streptococcus pyogenes. Methicillin-resistant Staphylococcus aureus (MRSA) has been a problem for many years in the hospital setting, more recently community acquired MRSA (CA-MRSA) has emerged posing additional challenges to physicians managing skin infection. The medicinal product under development, Lytixar™, is a synthetic antimicrobial peptidomimetic agent with a membrane lysing mode of action. Lytixar™ has demonstrated activity against several Gram-positive and Gram-negative bacteria in vitro. The compound appears to be equally effective against antibiotic-resistant species such as methicillin resistant Staphylococcus aureus (MRSA), vancomycin resistant Enterococci (VRE) and multi-resistant Pseudomonas isolates. The novel membrane lysing mode of action may result in a lower propensity to the development of resistance and to date Lytixar™ demonstrates no in vitro target-specific cross-resistance with other classes of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 65, inclusive.
* Diagnosis of uncomplicated, Gram-positive, skin infection. This may include patients with mild eczema/dermatoses such as atopic dermatitis.
* Gram-positive organisms determined at Baseline (Day 1) which in the opinion of the investigator are causative for infection of the lesion(s).

Candidate for treatment with topical antibacterial therapy:

* area to be treated ≤100 cm2
* SIRS score of at least 8 for the area of study medication application

  * Female patients of child bearing potential and male patients with female partners of child-bearing potential must be willing to use an adequate barrier form of contraception, (i.e., diaphragm or condom with spermicidal agent) prior to entry into the study and for two weeks following the completion of all follow-up procedures. Hormonal contraception or hormonal IUDs alone are not considered to be acceptable forms of contraception.
  * Provision of signed and dated written informed consent by the patient.
  * Patient's medical condition is stable, with no other clinically significant abnormalities as determined by the investigator.
  * Patients must be able to understand the written patient information and the consent form, and be willing to return to the study site for follow up visits, comply with requirements, instructions and restrictions of the study as listed in the informed consent form.

Exclusion Criteria:

* Moderate to Severe dermatoses including but not limited to psoriasis, atopic dermatitis or eczema.
* Secondarily-infected animal/human bite, puncture wound or abscess.
* Chronic ulcerative lesions.
* Bacterial skin infection which, due to the area, depth or severity, in the opinion of the investigator, cannot be appropriately treated by a topical antibiotic.
* More than one type of infected lesion.
* Surgical intervention is required for treatment of the infection prior to enrolment in the study, or such intervention is likely to be required during the course of the study.
* Application of any topical pharmaceutical agent (including but not limited to, corticosteroids, antibacterials, antiseptics or antifungal agents) directly to the infected wound/lesion(s), within 72 hours prior to study entry.
* Systemic signs or symptoms of infection (such as fever).
* Treatment for one or more days with a systemic antibacterial agent within 72 hours of study entry.
* Ongoing treatment with systemic corticosteroids at a dose of >0.125mg/kg per day of prednisone (or the equivalent).
* Known, pre-existing or serious underlying disease that could be imminently life-threatening.
* Pregnancy or ongoing lactation.
* Participation in any study using an investigational drug or device during the previous 30 days prior to entering the study.
* Significant ongoing or history of drug or alcohol abuse which in the opinion of the investigator makes the patient unsuitable for enrolment.
* Known allergic reactions or hypersensitivity of significant severity in general and specifically to any component of the study medication.
* Current or history of significant hepatic, renal, endocrine, cardiac, nervous, psychiatric, gastrointestinal, pulmonary, haematological, or metabolic disorder that is not in a stable condition. Malignancy <5 years since last treatment (resolved basal cell carcinoma is permitted).
* Current or history of any significant disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Other unspecified reasons that, in the opinion of the investigator make the Patient unsuitable for enrolment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To determine the safety and local tolerability of topically administered Lytixar™ in patients with uncomplicated, Gram-positive, skin infection. | After topical treatment 3 times per day 5 days
  Tolerability and safety will be measured at Day 3, the end of treatment visit Day 7 and follow-up visits Day 14, and 21.

SECONDARY OUTCOMES:
To assess the clinical and microbiological response to Lytixar™ in patients with uncomplicated, Gram-positive, skin infection. And to determine the extent of systemic absorption of Lytixar™. | Topical treatment 3 times daily for 5 days.
  Clinical outcome, changes in the Skin Infection Rating Scale (SIRS) scores from Baseline, and Bacteriological success, recurrence, failure or evaluability will be assessed at Day 3, end of treatment visit Day 7 and follow-up visits Day 14 and 21.

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Kemeny, DSc, Prof, Principal Investigator — St. George Albert Clinic Zeged University Hospital
Locations (4):
- Hungary (4):
  - Debreceni Egyetem Orvos-és Egészségtudományi, Debrecen
  - Miskolci Semmelweis Ignác Egészegügyi Központ és, Miskolc
  - Pécsi Tudományegyetem általános Orvostudom´nyi Centum, Pécs
  - Szeged Univesrity Hospital, Szeged